CLINICAL TRIAL: NCT00370747
Title: Efficacy and Safety of Ecabet Ophthalmic Solution for the Treatment of Dry Eye Syndrome
Brief Title: Efficacy and Safety Study for Ecabet Ophthalmic Solution for Treating Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISTA-ECBT-CS02
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — ecabet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ecabet (Experimental): Ophthalmic solution in the Study eye four times daily for 90 days.
  Interventions: Drug: Ecabet
- Placebo (Placebo Comparator): Ophthalmic solution in the Study eye four times daily for 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ecabet — ophthalmic solution 2.83%
  Arms: Ecabet
Drug: Ecabet — ophthalmic solution 3.70%
  Arms: Ecabet
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether ecabet ophthalmic solution is an effective treatment for dry eye syndrome

ELIGIBILITY:
Inclusion Criteria:

* Male/female at least 18 years of age
* Agree to avoid disallowed medications
* Have a diagnosis of dry eye

Exclusion Criteria:

* Have chronic systemic inflammation
* Have active seasonal ocular allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Ocular signs and Symptoms | 90 days
  ocular signs, including corneal and conjunctival staining, tear film breakup time and blink rate, and ocular symptoms, including burning or stinging, itchiness or scratchiness, grittiness or sandiness, foreign body sensation, haziness or blurriness, photophobia, photopsia, and eye discomfort

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | 90 days
  Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Bianca, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- Irvine, California, United States